CLINICAL TRIAL: NCT04657458
Title: Bone Marrow Mesenchymal Stem Cell Derived Extracellular Vesicles Infusion Treatment: Expanded Access Protocol for Patients With COVID-19 Associated ARDS
Brief Title: Expanded Access for Use of bmMSC-Derived Extracellular Vesicles in Patients With COVID-19 Associated ARDS
Status: No longer available | Type: Expanded Access
Sponsor: Direct Biologics, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: DB-EF-EXPANDEDACCESS-001
Record Dates: First submitted 2020-12-07; First posted 2020-12-08 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Covid19; ARDS; Hypoxia; Cytokine Storm
Keywords: COVID-19; ARDS; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Hypoxia; Cytokine Release Syndrome

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: ExoFlo — Intravenous administration of bone marrow mesenchymal stem cell derived extracellular vesicles

SUMMARY:
ExoFlo, Bone Marrow Mesenchymal Stem Cell Derived Extracellular Vesicles Allograft Product, Infusion Treatment is currently being studied in Protocol DB-EF-PhaseIII-0001 in patients COVID-19 associated moderate to severe acute respiratory distress syndrome (ARDS). This expanded access protocol is an open label study intended to provide ExoFlo to critically ill patients who do not qualify for the Phase III randomized controlled trial (RCT) because they

* Do not meet phase III eligibility criteria at current phase III sites.
* Do meet phase III eligibility criteria but cannot access phase III sites.
* Do not meet phase III eligibility criteria & cannot access phase III sites.

DETAILED DESCRIPTION:
Objectives:

First, to provide Investigational Medicinal Product (IMP) to patients with COVID-19 associated moderate to severe ARDS who do not qualify for Protocol DB-EF-PHASEIII-0001. Secondarily, to collect safety and efficacy data.

Endpoints:

Primary Endpoint:

1) 60-day All-Cause Mortality

Secondary Endpoints:

1. Incidence of serious adverse events (SAEs).
2. Ventilator-free days (VFDs).
3. Time to discharge.

Exploratory Endpoints:

1. Acute phase reactants: C-reactive protein (CRP), D-dimer, and Ferritin change from Baseline on Days 3, 5, 7, 10, 15, and 29 for subjects who are still hospitalized.
2. Sequential Organ Failure Assessment (SOFA) Score change from Baseline on Days 15, and 29 for subjects who are still hospitalized.
3. Improvement in partial pressure of arterial oxygen to fraction of inspired oxygen (PaO2/FiO2) ratio from pre-infusion baseline (Day 0) to Day 7. PaO2 may be calculated from arterial blood gas (ABG) or imputed from the SpO2 daily.

Number of subjects: ≤200

Phase: Phase II /Expanded Access Protocol for Intermediate Population

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent by self or proxy.
2. Stated willingness to comply with study protocol.
3. Male or female of any age ≥ 18 years of age
4. May be pregnant unless the patient has one or more conditions listed under Exclusion Criteria #3.
5. Positive Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) SARS-CoV-2.
6. Moderate to severe ARDS as defined by timing within ten days of known clinical insult or new or worsening respiratory symptoms, bilateral opacities not fully explained by effusions or lung collapse, and respiratory failure not fully explained by cardiac failure or fluid overload, minimum 5 cm H2O PEEP on mechanical ventilation, and PaO2/FiO2 ≤ 200 mmHg (if using an estimated P/F ratio, a S/F ≤ 235 is accepted).
7. Acute presentation of hypoxic respiratory failure requiring noninvasive oxygen support OR mechanical ventilation (MV).

Exclusion Criteria:

1. Active malignancy requiring treatment within the last two years, with the exception of non-melanoma skin cancers.
2. Patients who are not full code.
3. Pregnant patients with current or past history of eclampsia, preeclampsia, hemolysis, elevated liver enzymes, or low platelet count (HELLP) syndrome during pregnancy.
4. New York Heart Association (NYHA) Functional Class III (symptoms present during ordinary activities) or IV Heart Failure (symptoms present at rest) or listed for heart transplant.
5. Chronic Kidney Disease (CKD) Stage IV (GFR 15-29 mL/min/1.73m2) and Stage V (GFR < 15 mL/min/1.73m2) or listed for kidney transplant.
6. Hepatic Impairment with Model for End-Stage Liver Disease (MELD) score ≥ 30 or listed for liver transplant.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bill Arana, Study Director — Direct Biologics, LLC

REFERENCES:
- See also: Direct Biologics, LLC — https://directbiologics.com/